CLINICAL TRIAL: NCT06382948
Title: A Randomized Phase 3, Double-Blind, Placebo-Controlled Study of Elacestrant Plus Everolimus Versus Elacestrant in Patients With ER+/HER2-, ESR1mut Advanced Breast Cancer Progressing to Endocrine Therapy and CDK4/6 Inhibitors
Brief Title: Elacestrant + Everolimus in Patients ER+/HER2-, ESR1mut, Advanced Breast Cancer Progressing to ET and CDK4/6i.
Acronym: ADELA
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: MedSIR (Other)
Collaborators: Stemline Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MedOPP545; 2024-512926-27-00 (EU CTIS Number)
Record Dates: First submitted 2024-04-05; First posted 2024-04-24 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2024-12

CONDITIONS: Advanced Breast Cancer; ER-positive Breast Cancer; HER2-negative Breast Cancer; ESR1 Gene Mutation
Keywords: ER-positive; HER22-negative; ESR1-mutation; CDK4/6-inhibitor; Selective endocrine receptor degrader (SERD)
MeSH Terms: interventions — Everolimus; elacestrant; RAD1901; Selective Estrogen Receptor Modulators; Gonadotropin-Releasing Hormone

STUDY DESIGN:
Intervention Model Description: Double-blind, parallel group (two arms: elacestrant plus everolimus, and elacestrant plus placebo).
Who Masked: Participant, Investigator
Masking Description: A blinded, independent IRC will perform a review of radiographic images and clinical information collected on study to determine the protocol-defined endpoints of disease response and progression. Further information on the independent review process will be provided in the BIRC Charter.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interventional Arm 1 (Experimental): Patients will receive 345 mg of elacestrant and 7.5 mg of everolimus orally once daily.
  Patients will remain in treatment until disease progression, treatment discontinuation, the start of new anti-cancer treatment, withdrawal of consent, death, or EoS, whichever occurs first.
  Interventions: Drug: Everolimus; Drug: Elacestrant; Drug: Auxiliary Medicinal Product - Dexamethasone; Drug: Auxiliary Medicinal Product - Luteinizing hormone-releasing hormone (LHRH) analogues
- Control Arm 2 (Active Comparator): Patients will receive elacestrant at (345 mg orally once daily) plus matched everolimus placebo.
  Patients will remain in treatment until disease progression, treatment discontinuation, the start of new anti-cancer treatment, withdrawal of consent, death, or EoS, whichever occurs first.
  Interventions: Drug: Elacestrant; Drug: Placebo; Drug: Auxiliary Medicinal Product - Dexamethasone; Drug: Auxiliary Medicinal Product - Luteinizing hormone-releasing hormone (LHRH) analogues

INTERVENTIONS:
Drug: Everolimus — Patients will receive 7.5 mg of everolimus orally once daily.
  Other Names: Zortress; Votubia; RAD001; Certican; Afinitor
  Arms: Interventional Arm 1
Drug: Elacestrant — Patients will receive elacestrant 345 mg orally once daily
  Other Names: ER-306323; RAD1901; Selective estrogen receptor degrader/selective estrogen receptor modulator (SERD/SERM) RAD1901
Drug: Placebo — Patients will receive placebo orally once daily
  Arms: Control Arm 2
Drug: Auxiliary Medicinal Product - Dexamethasone — 10 mL of alcohol-free dexamethasone 0.5 mg per 5 mL mouthwashes (swish for 2 min and spit, four times daily for 8 weeks). After 8 weeks, dexamethasone mouthwash could be continued for up to eight additional weeks at the discretion of the clinician and patient. Used for prevention of treatment-induced stomatitis.
Drug: Auxiliary Medicinal Product - Luteinizing hormone-releasing hormone (LHRH) analogues — According to clinical practice (for premenopausal/perimenopausal patients and male patients in both treatment arms). Used to suppress estrogen production.

SUMMARY:
This trial will study a type of advanced breast cancer (ABC) defined as endocrine receptor (ER)-positive/human epidermal growth factor receptor 2(HER2)-negative and estrogen receptor 1 (ESR1)-mutated. Patients will be treated with elacestrant, a compound that acts as a selective estrogen receptor degrader, and everolimus (or placebo), a kinase inhibitor indicated for the treatment of postmenopausal women with advanced hormone receptor-positive, HER2-negative breast cancer.

The main purpose of the study is to analyze the efficacy (to find out how effective a treatment is) of elacestrant plus everolimus therapy in patients who have ER-positive/HER2-negative, ESR1-mutated, ABC progressing to endocrine therapy and cyclin-dependent kinase 4/6 (CDK4/6) inhibitor. The efficacy of elacestrant plus everolimus combination will be determined by assessing the period from elacestrant plus everolimus (or placebo) treatment initiation until to the first occurrence of disease progression, unacceptable toxicity, death, or discontinuation from the study treatment for any other reason, whichever occurs first, defined as progression free survival.

Rigorous eligibility criteria based on specific co-morbidities and clinicopathologic features of their disease have been designed to minimize the risk of patients participating in this study. The anticipated favorable clinical benefits of elacestrant combined with everolimus are projected to outweigh the risks of this treatment. This study will be performed in full compliance with International Council for Harmonisation of Technical Requirements for Pharmaceuticals for Human Use (ICH) and all applicable local Good Clinical Practice (GCP) and regulations.

DETAILED DESCRIPTION:
Upon meeting all selection criteria, a total of 240 patients will be enrolled.

After signing the Informed Consent Form (ICF), patients will be randomized (ratio 1:1) as follows:

* Interventional Arm (Arm A) (N=120): Patients will receive 345 mg of elacestrant and 7.5 mg of everolimus orally once daily.
* Control Arm (Arm B) (N=120): Patients will receive elacestrant at 345 mg orally once daily plus everolimus placebo.

Patients will be stratified by presence of visceral metastases (yes versus no) and duration of prior CDK4/6 inhibitor-based therapy (≥ 12 months versus < 12 months). Patients progressing to CDK4/6 inhibitor-based therapy in the adjuvant setting will be stratified as patients with a duration of prior CDK4/6 inhibitor-based therapy < 12 months.

Patients will receive study treatment in 28-day cycles until documented disease progression, death, unacceptable toxicity, or discontinuation from the study treatment for any other reason, whichever occurs first.

Patients discontinuing the study treatment period will enter a post-treatment follow-up period during which survival and new anti-cancer therapy information will be collected every 3 months (± 14 days) from the last dose of IMPs until the End of Study (EoS) defined as 12 months after last patient is randomized unless premature termination of the trial. For patients who discontinue the study treatment for reasons other than disease progression, tumor assessments will be conducted following the frequency of the study until the start of a new anti-cancer treatment, death, or disease progression.

ELIGIBILITY:
Inclusion Criteria:

Patients will be included in the study only if they meet ALL of the following criteria:

1. Patient must be capable to understand the purpose of the study and have signed written informed consent form (ICF) prior to beginning specific protocol procedures.
2. Female or male patients ≥ 18 years of age at the time of signing ICF.
3. Pre- or perimenopausal women, who do not meet the criteria for post-menopausal status (defined in continuation) and men must be concurrently receiving a LHRH analogue for at least 28 days (if shorter, post-menopausal levels of serum estradiol/follicle-stimulating hormone [FSH] must be confirmed analytically) prior to study randomization and are planning to continue LHRH agonist treatment during the study.

   Post-menopausal women as defined by any of the following criteria:
   1. Age ≥ 60 years;
   2. Age < 60 years and cessation of regular menses for at least 12 consecutive months with no alternative pathological or physiological cause; and serum estradiol and/or FSH levels within the laboratory's reference range for post-menopausal females;
   3. Documented bilateral surgical oophorectomy.
4. Histologically- or cytologically proven diagnosis of adenocarcinoma of the breast with evidence of either unresectable locally recurrent or metastatic disease confirmed by computerized tomography (CT) scan or magnetic resonance imaging (MRI) that is not amenable to resection with curative intent.
5. Documentation of ER[+] (≥10% positive stained cells) and HER2[-] (0-1+ by immunohistochemistry [IHC] or 2+ and negative by in situ hybridization [ISH] test) tumor according to the most recent American Society of Clinical Oncology (ASCO)/College of American Pathologists (CAP) guidelines as per local assessment. ER[+]/HER2[-] status should be confirmed in metastatic setting, with exception of patients with bone and lung only disease.
6. Patients with ESR1 mutational status will be determined before patient randomization using Guardant360 CDx (Guardant Health) test.

   Note: Patients with previously determined ESR1 mutation using appropriately validated tests (Guardant360 CDx [Guardant Health], FoundationOne CDx, FoundationOne Liquid [Foundation Medicine Inc]) will be eligible for inclusion. This local determination can be performed either in blood or tumor samples.
7. Radiological or objective evidence of disease progression on prior treatment with a CDK4/6 inhibitor in combination with endocrine therapy for advanced disease after at least 6 months of treatment. Patients receiving CDK4/6 inhibitor-based therapy in the adjuvant setting are also eligible provided that disease progression is confirmed after at least 12 months of treatment but no more than 12 months following CDK4/6 inhibitor treatment completion in this scenario.
8. Patients must have previously received at least one and no more than two lines of endocrine therapy for ABC. Progression during or within 12 months of adjuvant endocrine therapy is considered as a line of endocrine therapy for advanced disease.
9. No prior elacestrant or other investigational SERDs, proteolysis targeting chimera (PROTAC), complete estrogen receptor antagonist (CERAN), or novel SERM, and/or PI3K/AKT/mTOR inhibitors, including everolimus, for advanced disease are permitted.

   Note: Fulvestrant is permitted if treatment was completed administered at least 28 days before randomization.
10. No prior chemotherapy for advanced disease is allowed.
11. Evidence of measurable disease as per Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v.1.1), or non-measurable, but evaluable, disease, including bone-only disease with at least one lytic or mixed lytic-blastic bone lesion.
12. Willingness and ability to provide the most recently available formalin-fixed paraffin-embedded (FFPE) tumor tissue or block. If a newly obtained baseline biopsy of an accessible tumor lesion is not possible to be obtained prior randomization, an archival tissue sample will be accepted.
13. Fasting serum cholesterol ≤ 300 mg/dL or 7.75 mmol/L and fasting triglycerides ≤ 2.5 times the upper limit of normal (x ULN).
14. Adequate bone marrow and organ function:

    1. Hematological (without platelet, red blood cell transfusion, and/or granulocyte colony-stimulating factor support within seven days before randomization): absolute neutrophil count (ANC) ≥ 1.5 x 109/L; platelet count ≥ 100.0 x109/L; and hemoglobin ≥ 9.0 g/dL.
    2. Hepatic: Serum albumin ≥ 2.5 g/dL; total serum bilirubin < 1.5 x ULN except for patients with Gilbert's syndrome who may be included if the total serum bilirubin is ≤ 3 x ULN or direct bilirubin ≤ 1.5 x ULN; alkaline phosphatase (ALP) ≤ 2.5 x ULN (≤ 3 x ULN in patients with liver and/or bone metastases); aspartate transaminase (AST) and alanine transaminase (ALT) ≤ 1.5 x ULN (≤ 3 x ULN in patients with liver metastases).
    3. Renal: Serum creatinine ≤ 1.5 x ULN or estimated creatinine clearance ≥ 50 mL/min as calculated by Cockcroft- Gault equation.
    4. Coagulation: International normalized ratio (INR) ≤ 1.5 x ULN, unless that the patient meets the exception described in the exclusion criteria 16.
15. Resolution of all acute toxic effects of prior anti-cancer therapy to grade ≤ 1 as determined by the National Cancer Institute (NCI)-Common Terminology Criteria for Adverse Events (CTCAE) v.5.0 (except for toxicities not considered a safety risk for the patient at Investigator's discretion).

    Note: Patients with grade 2 alopecia are allowed.
16. Women of childbearing potential who are sexually active with a non-sterilized male partner must have a negative serum pregnancy test within 7 days before randomization. In addition, they agree to use one highly effective method of birth control 28 days prior to start of treatment until 120 days after the last dose of study treatments. Female patients must refrain from egg cell donation and breastfeeding during this same time period.
17. Male participants with a female partner of childbearing potential must be surgically sterile or using a highly effective method of contraception 28 days prior to treatment until 120 days after the last dose of study treatments to prevent pregnancy in a partner. Male participants must not donate or bank sperm during this same time period. Not engaging in heterosexual activity (sexual abstinence) for the duration of the study and 120 days after the last dose of study treatments is an acceptable practice if this is the preferred usual lifestyle of the participant.
18. ECOG performance status of 0-1.
19. Minimum life expectancy of ≥ 12 weeks at screening.

Exclusion Criteria:

Any patient meeting ANY of the following criteria will be excluded from the study:

1. Inability to comply with study and follow-up procedures.
2. Formal contraindication to endocrine therapy defined as visceral crisis and/or rapidly or symptomatic progressive visceral disease.
3. Current participation in another therapeutic clinical trial.
4. Treatment with approved or investigational cancer therapy within 14 days prior to randomization except for fulvestrant that must be administered completed at least 28 days before randomization.
5. Known active uncontrolled or symptomatic central nervous system (CNS) metastases and/or leptomeningeal disease as indicated by clinical symptoms, cerebral edema, and/or progressive growth. Patients with a history of CNS metastases are eligible if they have been previously treated with local therapy, are clinically stable, and off anticonvulsants and steroids for at least 14 days before randomization.
6. Intact uterus with a history of endometrial intraepithelial neoplasia (atypical endometrial hyperplasia or higher-grade lesion).
7. Concurrent malignancy or malignancy within three years before randomization with the exception of carcinoma in situ of the cervix, non-melanoma skin carcinoma, or stage I uterine cancer. For other cancers considered to have a low risk of recurrence, discussion with the Medical Monitor is required.
8. Known allergy or hypersensitivity reaction to any investigational medicinal products (IMPs) or their incorporated substances.
9. History of malabsorption syndrome or other condition that would interfere with enteral absorption (ongoing gastrointestinal obstruction/motility disorder, malabsorption syndrome, or prior gastric bypass) or results in the inability or unwillingness to swallow pills.
10. Palliative radiotherapy with a limited field of radiation within two weeks or with wide field of radiation or to more than 30% of the bone marrow within four weeks prior to randomization.
11. Major surgical procedure or significant traumatic injury within 14 days before randomization or anticipation of need for major surgery within the course of the study treatment.
12. Clinically relevant cardiovascular/cerebrovascular disease and/or cardiac dysfunction or conduction abnormalities including, but not confined, to any of the following:

    a. Symptomatic pericarditis, unstable angina pectoris, documented myocardial infarction, coronary/peripheral artery bypass graft, symptomatic cardiac heart failure (CHF) (New York Heart Association [NYHA] Class II-IV), or cerebrovascular accident including transient ischemic attack within six months before study randomization.
13. Concurrent uncontrolled atrial fibrillation, other ongoing cardiac dysrhythmias grade ≥ 2 as determined by NCI-CTCAE v.5.0, or prolonged QT Interval Corrected by Fridericia's formula ([QTcF] > 480 msec).
14. Clinically severe pulmonary compromise resulting from intercurrent pulmonary illnesses including, but not limited, to any of the following:

    1. Massive lung metastatic involvement (e.g., pleural effusion, lymphangitic carcinomatosis, etc.).
    2. Any underlying pulmonary disorder (e.g., severe asthma, severe chronic obstructive pulmonary disease [COPD], restrictive lung disease, post Coronavirus disease (COVID-19) pulmonary fibrosis, etc.).
    3. Any autoimmune, connective tissue, or inflammatory disorders with pulmonary involvement (e.g., rheumatoid arthritis, Sjogren's syndrome, sarcoidosis, etc.).
    4. Prior pneumonectomy.
15. History of non-infectious interstitial lung disease (ILD)/pneumonitis that required steroids, has current ILD/pneumonitis, or has suspected ILD/pneumonitis that cannot be ruled out by imaging at screening.
16. Coagulopathy or any history of coagulopathy within six months before study enrollment, including history of deep vein thrombosis or pulmonary embolism. However, patients with the following conditions will be allowed to participate:

    1. Adequately treated catheter-related venous thrombosis occurring more than 28 days prior to randomization.
    2. Treatment with an anticoagulant (e.g., warfarin or heparin) for a thrombotic event occurring more than six months before randomization, or for an otherwise stable and allowed medical condition (e.g., well controlled atrial fibrillation), provided dose and coagulation parameters (as defined by local standard of care) are stable for at least 28 days prior to randomization.
17. Concomitant treatment with immunosuppressive agents or chronic corticosteroids use before randomization with the following exceptions: topical applications, inhaled sprays, eye drops, mouthwash, or local injections are allowed. Patients on stable low dose of corticosteroids ( ≤ 10 mg/day of prednisone or equivalent) for at least two weeks before randomization are also permitted.
18. Unable or unwilling to avoid prescription medications, over-the-counter medications, dietary/herbal supplements (e.g., St. John's wort), and/or foods (e.g., grapefruit, pomelos, star fruit, Seville oranges and their juices) that are moderate/strong inhibitors or inducers of CYP3A4 activity. Participation will be allowed if the medication, supplements, and/or foods are discontinued for at least five half-lives or 14 days (whichever is shorter) prior to randomization and for the duration of the study.
19. Pregnant or lactating women or patients not willing to apply highly effective contraception as defined in the protocol.
20. Current known infection with human immunodeficiency virus (HIV), hepatitis B virus (HBV), or hepatitis C virus (HCV). Patients with past HBV infection or resolved HBV infection (defined as having a negative hepatitis B surface antibody [HBsAg] test and a positive hepatitis B core antibody [HBcAb] test, accompanied by a negative HBV DNA test) are eligible. Patients positive for HCV antibody are eligible only if polymerase chain reaction (PCR) is negative for HCV RNA. Any other active uncontrolled infection at the time of screening is not allowed.
21. Known substance abuse or any other concurrent severe and/or uncontrolled psychiatric or medical condition that would, in the Investigator's judgment, contraindicate patient participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2024-12-05 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2028-04 (Estimated)

PRIMARY OUTCOMES:
To demonstrate superiority of elacestrant+everolimus vs. elacestrant+placebo in prolonging PFS based on a BIRC in patients with ER[+]/HER2[-], ESR1-mutated, ABC that have previously received ET+CDK4/6i (all patients). | Until disease progression, treatment discontinuation, the start of new anti-cancer treatment, withdrawal of consent, death, or EoS, whichever occurs first, assessed through study completion, an average of 12 months.
  Progression Free Survival (PFS), defined as the period from randomization to the first occurrence of disease progression or death from any cause, whichever occurs first, as assessed by a Blinded Imaging Review Committee (BIRC) through the use of RECIST v.1.1.

SECONDARY OUTCOMES:
To compare overall survival (OS) between treatment groups, in all patients. | Until disease progression, treatment discontinuation, the start of new anti-cancer treatment, withdrawal of consent, death, or EoS, whichever occurs first, assessed through study completion, an average of 12 months.
  OS, defined as the period from randomization to death from any cause, as determined locally by the Investigator.
To compare investigator-assessed PFS based on local assessment between treatment groups, in all patients. | Until disease progression, treatment discontinuation, the start of new anti-cancer treatment, withdrawal of consent, death, or EoS, whichever occurs first, assessed through study completion, an average of 12 months.
  Investigator-assessed PFS, defined as the period from randomization to the first occurrence of disease progression or death from any cause, whichever occurs first, as determined locally using RECIST v.1.1.
To compare objective response rate (ORR) between treatment groups, in all patients. | Until disease progression, treatment discontinuation, the start of new anti-cancer treatment, withdrawal of consent, death, or EoS, whichever occurs first, assessed through study completion, an average of 12 months.
  ORR is defined as the rate of patients with a Best Overall Response (BOR) of complete response (CR) or partial response (PR) based on a BIRC and local Investigator assessment through the use of RECIST v.1.1.
To compare clinical benefit rate (CBR) between treatment groups, in all patients. | Until disease progression, treatment discontinuation, the start of new anti-cancer treatment, withdrawal of consent, death, or EoS, whichever occurs first, assessed through study completion, an average of 12 months.
  CBR is defined as the rate of patients with an objective response (CR or PR), or stable disease for at least 24 weeks based on a BIRC and local Investigator assessment through the use of RECIST v.1.1.
To compare overall time to response (TTR) between treatment groups, in all patients. | Until disease progression, treatment discontinuation, the start of new anti-cancer treatment, withdrawal of consent, death, or EoS, whichever occurs first, assessed through study completion, an average of 12 months.
  TTR is defined as the period from the randomization to time of the first objective tumor response (tumor shrinkage of ≥ 30%) observed for patients who achieved a BOR of CR or PR based on a BIRC and local Investigator assessment through the use of RECIST v.1.1.
To compare duration of response (DoR) between treatment groups, in all patients. | Until disease progression, treatment discontinuation, the start of new anti-cancer treatment, withdrawal of consent, death, or EoS, whichever occurs first, assessed through study completion, an average of 12 months.
  DoR is defined as the period from the first occurrence of a documented objective response to disease progression or death from any cause, whichever occurs first, based on a BIRC and local Investigator assessment through the use of RECIST v.1.1.
To compare best percentage of change in tumor burden between treatment groups, in all patients. | Until disease progression, treatment discontinuation, the start of new anti-cancer treatment, withdrawal of consent, death, or EoS, whichever occurs first, assessed through study completion, an average of 12 months.
  Best percentage of change from baseline in the size of target tumor lesions is defined as the biggest decrease, or smallest increase if no decrease will be observed, based on a BIRC and local Investigator assessment through the use of RECIST v.1.1.
To describe the changes in health-related quality-of-life (HRQoL) from baseline using the EuroQoL 5 Dimension 5 Level (EQ-5D-5L) scale. | Until disease progression, treatment discontinuation, the start of new anti-cancer treatment, withdrawal of consent, death, or EoS, whichever occurs first, assessed through study completion, an average of 12 months.
  Changes from baseline in the EQ-5D-5L scale. The descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels, indicating, from 1 to 5: no problems, slight problems, moderate problems, severe problems and extreme problems. The patient is asked to indicate their health state by ticking the box next to the most appropriate statement in each of the five dimensions. This decision results in a 1-digit number that expresses the level selected for that dimension. The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state.
To describe the changes in HRQoL from baseline using the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ-C30). | Until disease progression, treatment discontinuation, the start of new anti-cancer treatment, withdrawal of consent, death, or EoS, whichever occurs first, assessed through study completion, an average of 12 months.
  Changes from baseline in the EORTC QLQ-C30 scale. All of the scales and single item measures range in score from 0 to 100. A high score for the functional scales and functional single items represents a high/healthy level of functioning, whereas a high score for the symptom scales and symptom item represents a high level of symptomatology or problems.
To describe the changes in HRQoL from baseline using the EORTC Quality of Life Questionnaire Breast Cancer module (EORTC QLQ-BR42). | Until disease progression, treatment discontinuation, the start of new anti-cancer treatment, withdrawal of consent, death, or EoS, whichever occurs first, assessed through study completion, an average of 12 months.
  Changes from baseline in the QLQ-BR42 scale. All of the scales and single item measures range in score from 0 to 100. A high score for the functional scales and functional single items represents a high/healthy level of functioning, whereas a high score for the symptom scales and symptom item represents a high level of symptomatology or problems.
To assess adverse events (AEs) between treatment groups in all patients. | Until disease progression, treatment discontinuation, the start of new anti-cancer treatment, withdrawal of consent, death, or EoS, whichever occurs first, assessed through study completion, an average of 12 months.
  Measures will include AEs and treatment-emergent AEs (TEAEs), including NCI CTCAE v5.0 severity grade and relationship to study drugs.
To assess adverse events leading to study treatment withdrawal. | Until disease progression, treatment discontinuation, the start of new anti-cancer treatment, withdrawal of consent, death, or EoS, whichever occurs first, assessed through study completion, an average of 12 months.
  Measures will include deaths, serious adverse events (SAEs), and AEs leading to study treatment withdrawal.
To assess adverse events leading to dose modification. | Until disease progression, treatment discontinuation, the start of new anti-cancer treatment, withdrawal of consent, death, or EoS, whichever occurs first, assessed through study completion, an average of 12 months.
  Measures will include dose interruption and reductions due to AEs.
To assess the number of participants with abnormal hematology and/or chemistry values that are related to treatment. | Until disease progression, treatment discontinuation, the start of new anti-cancer treatment, withdrawal of consent, death, or EoS, whichever occurs first, assessed through study completion, an average of 12 months.
  Number of participants with treatment-related AEs as measured by laboratory parameters (hematology and chemistry) and assessed by NCI CTCAE v5.0 grade.
To assess the number of participants with changes on vital signs and/or AEs that are related to treatment. | Until disease progression, treatment discontinuation, the start of new anti-cancer treatment, withdrawal of consent, death, or EoS, whichever occurs first, assessed through study completion, an average of 12 months.
  Number of participants with treatment-related changes on vital sign values as determined by respiratory rate, blood pressure (systolic and diastolic), pulse rate, and body temperature over time and assessed by NCI-CTCAE v.5.0.
To assess the number of participants with changes on cardiac function measured by ECG QT Interval Corrected by Fridericia formula (QTcF) that are related to treatment effect . | Until disease progression, treatment discontinuation, the start of new anti-cancer treatment, withdrawal of consent, death, or EoS, whichever occurs first, assessed through study completion, an average of 12 months.
  Measurement of treatment-related changes in cardiac function measured by ECG QTcF over time.
To assess the number of participants with changes on Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) that are related to treatment. | Until disease progression, treatment discontinuation, the start of new anti-cancer treatment, withdrawal of consent, death, or EoS, whichever occurs first, assessed through study completion, an average of 12 months.
  Measurement of treatment-related changes on patient's level of functioning in terms of their ability to care for themself, daily activity, and physical ability (walking, working, etc.), as measured with the ECOG PS scale over time.

OTHER OUTCOMES:
Exploratory endpoint: protein expression studies using blood samples to investigate the potential association with clinical outcomes. | Until disease progression, treatment discontinuation, the start of new anti-cancer treatment, withdrawal of consent, death, or EoS, whichever occurs first, assessed through study completion, an average of 12 months.
  Protein expression (IHC and proteomics) profiling analyses performed on blood samples to investigate the potential association with clinical outcomes.
Exploratory endpoint: analysis of allele mutation frequencies in circulating tumor DNA (ctDNA) in blood samples to investigate the potential association with clinical outcomes. | Until disease progression, treatment discontinuation, the start of new anti-cancer treatment, withdrawal of consent, death, or EoS, whichever occurs first, assessed through study completion, an average of 12 months.
  Changes in biomarkers allele mutation frequencies in ctDNA in blood samples to investigate the potential association with clinical outcomes.
Exploratory endpoint: Genetic studies using blood samples to investigate the potential association with clinical outcomes. | Until disease progression, treatment discontinuation, the start of new anti-cancer treatment, withdrawal of consent, death, or EoS, whichever occurs first, assessed through study completion, an average of 12 months.
  Gene expression profiling analyses performed on blood samples to investigate the potential association with clinical outcomes.
Exploratory endpoint: Analysis of medical imaging (radiomics) to identify potential biomarkers associated with clinical outcomes. | Until disease progression, treatment discontinuation, the start of new anti-cancer treatment, withdrawal of consent, death, or EoS, whichever occurs first, assessed through study completion, an average of 12 months.
  Analysis of oncological biomarkers, such as growth rate of tumor derived by tumor growth rate modeling or tumor heterogeneity according to quantitative estimation performed on radiological images (radiomics) to investigate the potential association with clinical outcomes.
Exploratory endpoint: Pharmacokinetic (PK) parameter of maximum (Peak) Observed Serum Concentration (Cmax). | Until disease progression, treatment discontinuation, the start of new anti-cancer treatment, withdrawal of consent, death, or EoS, whichever occurs first, assessed through study completion, an average of 12 months.
  Blood samples of 40 patients/arm will be collected for the determination of Maximum Serum Concentration (Cmax).
  Timeframe: samples will be collected in a subset of approximately 40 patients/arm at Cycle 1 Day 14 at pre-dose (within 1h prior to study drug administration) and between 2 and 6h post-dose. Trough concentrations (pre-dose within 1h prior to study drug administration) will be collected at Day 1 of Cycle 3 and Day 1 of the following cycles every 8 weeks (CXD1) in conjunction with tumor assessments when applicable. Additional blood samples (one timepoint) for PK analysis will be collected in case of significant AE or SAEs considered as potentially related to the study drug (the time of the last dose intake and the sampling time should be reported to allow the determination of the corresponding actual time after dose).
Exploratory endpoint: Pharmacokinetic (PK) parameter of Plasma Through Concentration (Ctrough). | Until disease progression, treatment discontinuation, the start of new anti-cancer treatment, withdrawal of consent, death, or EoS, whichever occurs first, assessed through study completion, an average of 12 months.
  Blood samples of 40 patients/arm will be collected for the determination of Minimum Concentration (Plasma trough concentration [Ctrough]).
  Timeframe: samples will be collected in a subset of approximately 40 patients/arm at Cycle 1 Day 14 at pre-dose (within 1h prior to study drug administration) and between 2 and 6h post-dose. Trough concentrations (pre-dose within 1h prior to study drug administration) will be collected at Day 1 of Cycle 3 and Day 1 of the following cycles every 8 weeks (CXD1) in conjunction with tumor assessments when applicable. Additional blood samples (one timepoint) for PK analysis will be collected in case of significant AE or SAEs considered as potentially related to the study drug (the time of the last dose intake and the sampling time should be reported to allow the determination of the corresponding actual time after dose).

CONTACTS AND LOCATIONS:
Overall Officials: Javier Cortés, M.D., Ph.D., Principal Investigator — IOB Institute of Oncology, Quironsalud Group, Madrid & Barcelona, Spain; Antonio Llombart-Cussac, M.D., Ph.D., Principal Investigator — Arnau de Vilanova Hospital, Valencia, Spain; José Pérez-García, M.D., Ph.D., Principal Investigator — International Breast Cancer Center, Barcelona, Spain
Locations (69):
- Austria (3):
  - Medizinische Universität Innsbruck, Innsbruck
  - Ordensklinikum Linz Barmherzige Schwestern, Linz
  - Ordination Priv.-Doz. Dr. Michael Hubalek, Schwaz
- Czechia (3):
  - Masaryk Memorial Cancer Institute, Brno
  - Multiscan Nemocnice Horovice, Hořovice
  - Tomas Bata Regional Hospital in Zlin, Zlín
- France (7):
  - Polyclinique Bordeaux Nord Aquitaine, Bordeau
  - Centre Georges François Leclerc, Dijon
  - CHU Lyon Sud, Lyon
  - Hospital prive des Cotes d'Amor, Plérin
  - CHU Saint Etienne, Saint-Priest-en-Jarez
  - IUCT Oncopole, Toulouse
  - Institute de Cancerologie de Lorraine - Nancy, Vandœuvre-lès-Nancy
- Germany (2):
  - MVZ II der Niels Stensen Kliniken, Georgsmarienhütte
  - Klinikum Worms - Frauenklinik, Worms
- Greece (9):
  - University General Hospital Alexandroupoli, Alexandroupoli
  - 251 Air Force General Hospital, Athens
  - Aretaeio Hospital, Athens
  - Attikon University Hospital, Athens
  - Metropolitan General Hospital 4th department, Athens
  - University General Hospital of Heraklion, Heraklion
  - University General Hospital of Larissa, Larissa
  - Metropolitan Hospital Greece 1st department, Piraeus
  - EU Interbalkan Medical Center, Thessaloniki
- Italy (3):
  - Ospedali Riuniti Livorno, Livorno
  - Instituto Europeo di Oncologia, Milan
  - Azienda Ospedaliero- Universitaria Maggiore Della Carita, Novara
- Spain (39):
  - Centro Oncológico de Galicia, A Coruña
  - Complejo Hospitalario Universitario de Santiago (CHUS), A Coruña
  - Hospital General Universitario Dr. Balmis (Alicante), Alicante
  - Hospital Universitario San Juan de Alicante, Alicante
  - Institut Català d' Oncologia Badalona (ICO), Badalona
  - Hospital Clínic i Provincial de Barcelona, Barcelona
  - Hospital del Mar, Barcelona
  - Hospital Universitari Dexeus, Barcelona
  - Hospital Universitari Vall D'Hebron, Barcelona
  - Hospital Universitario de Basurto, Bilbao
  - Hospital Universitario de Burgos, Burgos
  - Hospital Provincial de Castellón, Castellon
  - Hospital San Pedro de Alcántara, Cáceres
  - Hospital Universitario Clínico San Cecilio de Granada, Granada
  - Complejo Hospitalario de Jaén, Jaén
  - Hospital Universitario Insular de Gran Canaria, Las Palmas de Gran Canaria
  - Hospital Universitario de León, León
  - Hospital Universitario Arnau de Vilanova de Lleida, Lleida
  - Hospital Beata María Ana, Madrid
  - Hospital Universitario Doce de Octubre, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario Puerta de Hierro Majadahonda, Madrid
  - Hospital Universitario Ramón y Cajal, Madrid
  - Hospital Universitario Sanchinarro-START-CIOCC, Madrid
  - MD Anderson Cancer Center Madrid, Madrid
  - Hospital Clínico Universitario Virgen de la Arrixaca, Murcia
  - Hospital Universitari Son Espases, Palma de Mallorca
  - Hospitalario Universitario de Navarra, Pamplona
  - Hospital Universitario de Canarias, Santa Cruz de Tenerife
  - Hospital Quirónsalud Sagrado Corazón, Seville
  - Hospital Universitario Virgen del Rocío, Seville
  - Hospital Universitario Virgen Macarena, Seville
  - Hospital Universitari Sant Joan de Reus, Tarragona
  - Hospital Universitario Marqués de Valdecilla, Valdecilla
  - Consorci Hospital General Universitari de València, Valencia
  - Hospital Arnau de Vilanova de Valencia, Valencia
  - Hospital Clínico Universitario de Valencia, Valencia
  - Hospital Universitario La Ribera - Alzira, Valencia
  - Hospital Clínico Universitario Lozano Blesa, Zaragoza
- United Kingdom (3):
  - Barts Health NHS Trust, London
  - Royal Cornwall Hospital NHS Trust, Truro
  - Genesis Cancer Care UK, Waterlooville